CLINICAL TRIAL: NCT06894186
Title: Comparison of the Functional Properties of Two Injectable Materials in Posterior Teeth: Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nourhan elsayed, Principal investigator, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Restoring class II cavities
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Class II Dental Caries; Dental Caries; Injectable Composite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- beautiful flow plus x (Experimental): shofu's beauitifil flow plus x is advanced bioactive material with the adaptability of flowable composite and mechanical properities of hybird composite
  Interventions: Other: Gaenial universal injectable

INTERVENTIONS:
Other: Gaenial universal injectable — GC Gaenial universal injectable advanced injectable composite with nano sized filler that merge the adaptation of flowable composite and mechanical properties of hybird composite

SUMMARY:
Using two different injectable materials in class II cavities to compare functional properties

ELIGIBILITY:
Inclusion Criteria:

* 1-Adult patients (20-50) 2-Good oral hygiene Good oral hygiene (Plaque index ≤2 (Moderate accumulation with plaque in the sulcus)) 3-Patient approval 4-Absence of parafunctional habits and/or bruxism 5-No endodontic treatment or abscess 6- class II either mesial or distal (no MOD cavities)

Exclusion Criteria:

* 1. Systematic disease that may affect participation. 2. Xerostomic patients. 3. Bad oral hygiene (plaque index 2 or 3) 14 4. Heavy smokers 5. Patients undergoing or will start orthodontic treatment 6. Signs and symptoms of irreversible pulpitis.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | T1: 1week T2: 6months T3 12 months
1- fracture of restoration and retention 2- proximal contact poiont | T(Time) T1:1 week hours beasline T2: 6 months T3:12 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hancer Sarica S, Arslan S, Balkaya H. Comparison of the 2-year clinical performances of class II restorations using different restorative materials. Clin Oral Investig. 2025 Feb 13;29(2):128. doi: 10.1007/s00784-025-06207-6. PMID 39945899
- [Result] Elderiny HM, Khallaf YS, Akah MM, Hassanein OE. Clinical Evaluation of Bioactive Injectable Resin Composite vs Conventional Nanohybrid Composite in Posterior Restorations: An 18-Month Randomized Controlled Clinical Trial. J Contemp Dent Pract. 2024 Aug 1;25(8):794-802. doi: 10.5005/jp-journals-10024-3737. PMID 39653674
- [Result] Rajabi H, Denny M, Karagiannopoulos K, Petridis H. Comparison of Flexural Strength and Wear of Injectable, Flowable and Paste Composite Resins. Materials (Basel). 2024 Sep 27;17(19):4749. doi: 10.3390/ma17194749. PMID 39410319
- [Result] Neto CCL, das Neves AM, Arantes DC, Sa TCM, Yamauti M, de Magalhaes CS, Abreu LG, Moreira AN. Evaluation of the clinical performance of GIOMERs and comparison with other conventional restorative materials in permanent teeth: a systematic review and meta-analysis. Evid Based Dent. 2022 Aug 1. doi: 10.1038/s41432-022-0281-8. Online ahead of print. PMID 35915167
- [Result] Ozer F, Patel R, Yip J, Yakymiv O, Saleh N, Blatz MB. Five-year clinical performance of two fluoride-releasing giomer resin materials in occlusal restorations. J Esthet Restor Dent. 2022 Dec;34(8):1213-1220. doi: 10.1111/jerd.12948. Epub 2022 Aug 7. PMID 35934807
- [Result] Deepika U, Sahoo PK, Dash JK, Baliarsingh RR, Ray P, Sharma G. Clinical evaluation of bioactive resin-modified glass ionomer and giomer in restoring primary molars: A randomized, parallel-group, and split-mouth controlled clinical study. J Indian Soc Pedod Prev Dent. 2022 Jul-Sep;40(3):288-296. doi: 10.4103/jisppd.jisppd_139_22. PMID 36260470
- [Result] 2022. Flowable GIOMER Vs Conventional Flowable Composite For Retention And Prevention Of Caries Recurrence When Used As Sealants For Initially Demineralized Fissures. A Randomized Clinical Trial. Journal of Pharmaceutical Negative Results. (Nov. 2022), 3257 3263
- [Result] Badr C, Spagnuolo G, Amenta F, Khairallah C, Mahdi SS, Daher E, Battineni G, Baba NZ, Zogheib T, Qasim SSB, Daher T, Chintalapudi N, Zogheib CM. A Two-Year Comparative Evaluation of Clinical Performance of a Nanohybrid Composite Resin to a Flowable Composite Resin. J Funct Biomater. 2021 Sep 9;12(3):51. doi: 10.3390/jfb12030051. PMID 34564200
- [Result] Kitasako Y, Sadr A, Burrow MF, Tagami J. Thirty-six month clinical evaluation of a highly filled flowable composite for direct posterior restorations. Aust Dent J. 2016 Sep;61(3):366-73. doi: 10.1111/adj.12387. PMID 26573239
- [Result] Kramer N, Reinelt C, Frankenberger R. Ten-year Clinical Performance of Posterior Resin Composite Restorations. J Adhes Dent. 2015 Aug;17(5):433-41. doi: 10.3290/j.jad.a35010. PMID 26525008
- [Result] Bayraktar Y, Ercan E, Hamidi MM, Colak H. One-year clinical evaluation of different types of bulk-fill composites. J Investig Clin Dent. 2017 May;8(2). doi: 10.1111/jicd.12210. Epub 2016 Jan 22. PMID 26800647